CLINICAL TRIAL: NCT04876924
Title: A Phase 1, Randomized, Double-Blinded, Placebo-controlled, Single and Multiple-Ascending Dose Study of the Safety, Tolerability, Food Effect, Pharmacokinetics, and Pharmacodynamics of BBP-711 (ORF-229) in Healthy Adult Subjects
Brief Title: A Study of BBP-711 (ORF-229) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cantero Therapeutics, a BridgeBio company (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ORF-01-001
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- BBP-711 for SAD (Experimental): A single dose of BBP-711 will be administered orally.
  Interventions: Drug: BBP-711
- Placebo for SAD (Placebo Comparator): A single dose of matching placebo will be administered orally.
  Interventions: Drug: Placebo
- BBP-711 for MAD (Experimental): A dose of BBP-711 will be administered orally for multiple days.
  Interventions: Drug: BBP-711
- Placebo for MAD (Placebo Comparator): A dose of matching placebo will be administered orally for multiple days.
  Interventions: Drug: Placebo
- BBP-711 for SAD Food Effect (Experimental): A single dose of BBP-711 will be administered orally.
  Interventions: Drug: BBP-711
- Placebo for SAD Food Effect (Placebo Comparator): A single dose of matching placebo will be administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BBP-711 — BBP-711, oral suspension
  Arms: BBP-711 for MAD; BBP-711 for SAD; BBP-711 for SAD Food Effect
Drug: Placebo — Placebo matching BBP-711
  Arms: Placebo for MAD; Placebo for SAD; Placebo for SAD Food Effect

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of BBP-711 in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a single-center, two-part, randomized, double-blinded, placebo-controlled, ascending dose study of BBP-711 in healthy male and female adult volunteers. The purpose of this study is to evaluate the safety and tolerability of BBP-711 in healthy adult volunteers. Each volunteer will participate in the study for about 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female who is 18 to 65 years old,
* Weight >50 kg and ≤110 kg at Screening
* Body mass index (BMI) 20 to 32 kg/m2, inclusive, at Screening
* In generally good health
* Nonsmoker, or not using tobacco or nicotine-containing products for at least 6 months

Exclusion Criteria:

* Use of any over-the-counter medications, including herbals or routine vitamins or minerals, or other supplements, within 7 days before admission to the research center.
* Pregnant or breastfeeding
* eGFR <90 mL/minute
* Abnormal ECG
* Abnormal laboratory results
* Positive test result for HIV, Hepatitis B, Hepatitis C, or COVID-19
* History of substance dependency (alcohol or other drugs of abuse) in the last 2 years
* Use of study drug in any clinical trial within 30 days of admission to the research center, or in the active follow-up phase of another clinical trial involving study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to Day 20
  Incidence of Adverse Events (AEs)

SECONDARY OUTCOMES:
Pharmacokinetic Assessments: Cmax | Blood samples will be taken pre-dose up to Day 10 for SAD and pre-dose up to Day 20 for MAD
  Maximum observed plasma concentration (Cmax)
Pharmacokinetic Assessments: Cmin | Blood samples will be taken pre-dose up to Day 10 for SAD and pre-dose up to Day 20 for MAD
  Minimum observed plasma concentration (Cmin)
Pharmacokinetic Assessments: AUC | Blood samples will be taken pre-dose up to Day 10 for SAD and pre-dose up to Day 20 for MAD
  Area under the plasma concentration-time curve from 0 to last measurable concentration (AUC(0-last)) computed using the linear trapezoidal rule
Pharmacodynamic Assessment: Baseline plasma glycolate | Baseline
  Baseline plasma glycolate
Pharmacodynamic Assessment: Percentage change from baseline plasma glycolate | Blood samples will be taken pre-dose up to Day 10 for SAD and pre-dose up to Day 20 for MAD
  Percentage change from baseline plasma glycolate
Pharmacodynamic Assessment: Baseline 24 Hour urinary glycolate:creatinine ratio | Baseline
  Baseline 24 Hour urinary glycolate:creatinine ratio
Pharmacodynamic Assessment: Percentage change from baseline of 24 Hour urinary glycolate:creatinine ratio | Urine samples will be taken pre-dose up to Day 3 for SAD and pre-dose up to Day 7 for MAD
  Percentage change from baseline of 24 Hour urinary glycolate:creatinine ratio

CONTACTS AND LOCATIONS:
Overall Officials: Terry O'Reilly, MD, Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No